CLINICAL TRIAL: NCT00765323
Title: Phase III, Open-Label, Multicenter International Study to Evaluate the Efficacy and Safety of an Octreotide Implant vs. Sandostatin LAR Depot in Patients With Acromegaly
Brief Title: Efficacy and Safety Study of Octreotide Implant in Patients With Acromegaly
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IP107-001
Record Dates: First submitted 2008-09-30; First posted 2008-10-02 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-09

CONDITIONS: Acromegaly
Keywords: Octreotide; Sandostatin LAR; Growth hormone; IGF-1
MeSH Terms: conditions — Acromegaly | interventions — Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 84 mg octreotide implant for 6 months
  Interventions: Drug: Octreotide Implant
- 2 (Active Comparator): Injections of Sandostatin LAR Depot(20, 30, 40 mg) every 4 weeks
  Interventions: Drug: Sandostatin LAR Depot

INTERVENTIONS:
Drug: Octreotide Implant — 84 mg octreotide subcutaneous implant for 6 months
  Other Names: somatostatin analogue
  Arms: 1
Drug: Sandostatin LAR Depot — Injections of Sandostatin LAR (dose range ~10-40 mg every 28 days)
  Other Names: somatostatin analogue
  Arms: 2

SUMMARY:
Evaluate the efficacy, safety and tolerability of the octreotide implant in patients with acromegaly that were previously treated with octreotide depot.

DETAILED DESCRIPTION:
This study will be conducted in 3 phases: Screening, the Primary Treatment Phase (ie, Day 1 to Week 24), and the Extension Phase (Post Week 24 to Week 48). Primary efficacy and safety will be determined from the Primary Treatment Phase. Eligible patients will be randomized during the Primary Treatment Phase; in a 3 to 1 ratio to receive 6 months of open-label treatment with either the 84 mg octreotide implant or monthy Injections of S-LAR. Each patient in this study will return to the investigational center every 4 weeks; safety and efficacy assessments will be performed during these visits. All patients who complete the Primary Treatment Phase and who continue to meet eligibility criteria will be offered the opportunity to enter the Extension Phase; patients entering the Extension Phase will be treated with an octreotide implant for 6 months.During the Extension Phase, patients will return to the investigational center every 4 weeks; safety and efficacy assessments will be performed during these visits.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with acromegaly
* Confirmed diagnosis of a growth hormone-secreting tumor
* Received a stable dose of monthly octreotide depot injections for a minimum of 3 consecutive months immediately prior to screening
* Must show a response to octreotide treatment with documented laboratory results at the screening visits defined as follows: IGF-1 < 20% above the upper limit of normal age and sex-adjusted levels and GH ≤ 2.5 ng/mL

Exclusion Criteria:

* Patients with pituitary surgery less than 3 months prior to screening
* Uncontrolled diabetes defined as having a fasting glucose > 150 mg/dl and HbA1c >= 9%
* Symptomatic cholelithiasis
* Received pegvisomant, Lanreotide, or a dopamine agonist within 3 months of screening, or at any time during the trial
* Received radiotherapy for pituitary tumor or any radiotherapy above the neck at any time before Screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2008-09; Primary Completion 2011-02 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Efficacy based on IGF-1, GH, signs and symptoms scores, tumor size, QoL and Patient Treatment Assessments | 12 months

CONTACTS AND LOCATIONS:
Locations (47):
- United States (8):
  - Stanford University Medical Center - Stanford Hospitals and Clinics, Palo Alto, California
  - University of Colorado - Veterans Administration Medical Center - Endocrinology, Denver, Colorado
  - Galiz Research, Miami, Florida
  - The University of Illinois at Chicago, Chicago, Illinois
  - Sinai Hospital of Baltimore, Medicine - Div. of Endocrinology and Metabolism, Baltimore, Maryland
  - The Cleveland Clinic, Cleveland, Ohio
  - Oregon Health and Science University, Endocrinology, Portland, Oregon
  - Seattle Neuroscience Institute - Swedish Medical Center, Seattle, Washington
- Czechia (2):
  - 2. interni klinika fakultní nemocnice Hradec Králové, Hradec Králové
  - 3. interni klinika Vseobecne fakultni nemocnice, Prague
- Germany (8):
  - Charité Berlin, Campus Benjamin Franklin, Abteilung fϋr Endokrinologie, Diabetes und Ernährungsmedizin, Berlin
  - Universitätsklinikum zu Köln, Klinik und Poliklinik II Innnere, Cologne
  - Universitätsklinikum Erlangen, Medizinische Klinik 1, Gastroenterologie, Pneumologie und Endokrinologie, Erlangen
  - Klinikum der Johann Wolfgang Goethe-Universität, Medizinische Klinik 1, Endokrinologie, Frankfurt
  - Universitätsklinikum Hamburg-Eppendorf - Bereich Endokrinologie, Diabetologie und Adipositas, Hamburg
  - Universitätsklinikum Schleswig-Holstein, Medizinische Klinik 1, Lübeck
  - Klinik für Endokrinologie und Stoffwechselkrankheiten Otto-von-Guericke-Universität Magdeburg, Magdeburg
  - Klinikum der Philipps Universitaet Marburg Bereich Endokrinologie & Diabetologie, Marburg
- Hungary (3):
  - Semmelweis University, Faculty of Medicine, 2nd Department of Medicine, Budapest
  - University of Debrecen Medical and Health Science Center, Division of Endocrinology, Debrecen
  - University of Pécs, School of Medicine, 1st Department of Medicine, Pécs
- Poland (5):
  - Akademickie Centrum Kliniczne - Szpital Akademii Medycznej w Gdańsku, Gdansk
  - Szpital Kliniczny im. Heliodora Święcickiego Uniwersytetu Medycznego im. Karola Marcinkowskiego w Poznaniu, Poznan
  - Indywidualna Specjalistyczna Praktyka Lekarska Dr n. med. Grzegorz Kulig, Szczecin
  - Szpital Bielański im. Ks. Jerzego Popiełuszki SPZOZ, Warsaw
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 we Wrocławiu, Klinika Endokrynologii, Diabetologii i Leczenia Izotopami, Wroclaw
- Russia (15):
  - National Educational Institution of Additional Professional Education "St. Petersburg Medical Academy of Postgraduate Studies of Roszdrav", Saint Petersburg, Russian Federation
  - State Institution of Healthcare "Regional Clinical Hospital", Barnaul
  - State Intitution of Healthcare "Mark of Honour "Irkutsk Regional Clinical Hospital", Irkutsk
  - State Institution of Healthcare "Kemerovo State Clinical Hospital", Kemerovo
  - Regional State Institution of Healthcare "Regional State Hospital", Krasnoyarsk
  - Federal State Institution "Endocrinology Research Center of Rosmedtechnology", Moscow
  - State Educational Institution of High Professional Education "Moscow Medical Academy named after I.M. Sechenov of Federal Agency of Healthcare and Social Development", Moscow
  - State Institution Moscow Regional Scientific-Research Clinical Institute named after M.F. Vladimirsky, Moscow
  - State Institution of Healthcare "N. Novgorod Regional Clinical Hospital named after N.A. Semashko", Nizhny Novgorod
  - State Educational Institution of High Professional Education "Novosibirsk State medical Univeristy of Federal Agency of Healthcare and Social Development, Novosibirsk
  - State Educational Institution of High Professional Education "Perm State Medical Academy named after academician E.A.Vagner of Roszdrav", Perm
  - Federal State Institution "federal Center of Heart, Blood and Endocrinology named after V.A. Almazov of Rosmedtechnology", Saint Petersburg
  - Center "Diabetes", LLC, Samara
  - State Educational Institution of High Professional Education "Siberian State Medical University of Federal Agency of Healthcare and Social Development", Tomsk
  - Municipal Health Care Institution Clinical Hospital for Emergency Medical Care named after N.V. Solovyov, Yaroslavl
- Institute of Endocrinology, Belgrade, Serbia
- Slovakia (2):
  - Endotopmed s.r.o., Tehelná, Bratislava
  - Národný endokrinologický a diabetologický ústav, Lubocna
- Spain (3):
  - Hospital General Universitario de Alicante Endocrinología y Nutrición, Alicante
  - Hospital Universitario Gregorio Marañón Endocrinología y Nutrición, Madrid
  - Hospital Universitario la Fé Endocrinología y Nutrición, Valencia

REFERENCES:
- [Derived] Chieffo C, Cook D, Xiang Q, Frohman LA. Efficacy and safety of an octreotide implant in the treatment of patients with acromegaly. J Clin Endocrinol Metab. 2013 Oct;98(10):4047-54. doi: 10.1210/jc.2013-2262. Epub 2013 Aug 22. PMID 23969184